CLINICAL TRIAL: NCT02917915
Title: The CaNadian Standardized Pulmonary Rehabilitation Efficacy Trial
Acronym: CoNSPiRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: McGill University (Other); University of Toronto (Other); Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Michael Stickland, Michael Stickland, PhD, Assistant Professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00066560
Record Dates: First submitted 2016-09-23; First posted 2016-09-28 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Emphysema; Chronic Bronchitis; Pulmonary rehabilitation; Lung Diseases, Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic; Lung Diseases, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- New Canadian Standardized PR (Experimental): * Education Content: exercise, living well with chronic lung disease, breathing management, conserving energy, pulmonary medications, inhaler devices, integrating exercise in your life, management of respiratory infections, management of aggravating environmental factors, management of stress & anxiety, nutrition, leisure & travel, getting a good night's sleep, enjoying intimacy, living in a smoke-free environment, integrating long-term oxygen into your life, keeping a healthy lifestyle.
  * Delivery style: During group sessions patients engage in active, participatory-based learning of program content. Workbooks are available. During one-on-one interactions motivational communication style (asking for permission before providing information, using open questions, etc.) is used.
  Interventions: Other: Canadian Standardized PR
- Traditional PR (Active Comparator): * Education Content: Exercise, anatomy, pulmonary diseases, healthier breathing, pulmonary medications, pulmonary devices, exercise action plan, allergies & pulmonary function tests, health and air quality, healthier eating, travel, stress management & relaxation, tips to remember/summary of content.
  * Delivery style: During group sessions, patients engage in passive learning of program content delivered in a lecture-style approach. Patients also receive one-on-one education regarding: dyspnea management/pacing, inhaler technique, exercise maintenance.
  Interventions: Other: Traditional PR

INTERVENTIONS:
Other: Canadian Standardized PR — Patients attend pulmonary rehabilitation (PR) 3 days per week for 6 weeks or 2 days per week for 8 weeks. Patients receive 2 hours of exercise training (aerobic and resistance) and 1 hour of education designed to promote self-management. In this intervention patients will receive the New Canadian Standardized PR educational approach (experimental).
  Arms: New Canadian Standardized PR
Other: Traditional PR — Patients attend pulmonary rehabilitation (PR) 3 days per week for 6 weeks or 2 days per week for 8 weeks. Patients receive 2 hours of exercise training (aerobic and resistance) and 1 hour of education designed to promote self-management. In this intervention patients will receive the Traditional PR education approach (active comparator).
  Arms: Traditional PR

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a chronic lung disease primarily caused by smoking. Pulmonary rehabilitation (PR) is an evidence-based, interdisciplinary, and comprehensive intervention for COPD patients that includes patient assessment, exercise training, and self-management education to promote behavior changes. PR has been shown to be the most effective strategy to improve clinical health outcomes, and is now considered to be a standard of care intervention for individuals with COPD who remain symptomatic despite optimal drug therapies. Despite considerable evidence supporting the effectiveness of PR at enhancing clinical outcomes, it is unclear if PR influences the behaviors that promote COPD management (i.e., physical activity, medication adherence, self-managing exacerbations).

In collaboration with the local clinical staff as well as national colleagues and the Canadian Thoracic Society, a new national pulmonary rehabilitation program has been co-developed that is designed to increase physical activity, medication adherence, and skills to help manage chronic lung diseases. The new program aims to increase people's confidence and autonomy for performing disease-management behaviors, and has been designed to be more effective at increasing physical activity, medication adherence, and disease management skills than previous pulmonary rehabilitation programs. The program is designed to be delivered within different settings of practice, including traditional PR centers, satellite sites (i.e., sites that are remote from the major institutions),with the use of Tele-health and web-based resources, and primary care medical centers. The effectiveness of the new Standardized Canadian PR program will be assessed relative to the traditional PR program. This trial is an important step towards establishing the necessary evidence that will then enable us to work on dissemination and implementation of this new standardized PR program across the country.

DETAILED DESCRIPTION:
Phase 1: The implementation of the new Canadian Standardized PR program "Real life project" will be done after evaluating the existing pulmonary rehabilitation program in each of the four sites (G.F. MacDonald Centre for Lung Health, Mount Sinai Hospital, Montreal Chest Institute and West Park Health Care Centre). This will serve as pilot testing of the new pulmonary rehabilitation program to identify problems, adapt solution and improve the program, its content and delivery.

Phase 2: A randomized parallel-controlled trial (RPCT) will also be implemented in one site at the G.F. MacDonald Centre for Lung Health. Entire PR classes will be block randomized according to a random numbers table to receive usual care (traditional PR) or the new Canadian Standardized PR program. Several rural Tele-health sites that participate in PR via the G.F. MacDonald Centre for Lung Health will also be included and randomized as well. Both groups will be exposed to the same exercise training component. The two groups will be exposed to different education components (described in detail elsewhere). The effectiveness of the new Canadian Standardized PR program (experimental group) will be evaluated relative to the Traditional PR program (active comparator group) in terms of clinical, behavioural, and psychological outcomes.

Primary Objective: To determine if the new Canadian Standardized PR program delivered in-person and in satellites sites with the support of Tele-health improves and maintains specific self-management behaviors after rehabilitation more than the traditional PR program.

Primary Outcome: Physical activity (in steps-per day as measured by Fitbit®) Secondary Outcomes: i) Medication adherence (measured by pharmacy refills); ii) exacerbation recognition and prompt decision-making (diary & phone calls).

Secondary Objectives: To determine if the new Canadian Standardized PR program improves predisposing factors of behavior change (knowledge, self-determination theory constructs such as motivation, and self-efficacy) following rehabilitation more than the Traditional PR program and if there is variation according to the method of delivering the program, i.e., via Tele-health technology vs in person.

To determine if the new Canadian Standardized PR program results in greater improvement of clinical outcomes (exercise capacity, health status) and health service use (hospital admissions) following completion of rehabilitation compared to the Traditional PR program.

Statistical Methods: Analysis for determining the potential benefit of the new Canadian Standardized PR program: Repeated measures ANOVAS will be conducted to evaluate changes over PR in behavioral outcomes (physical activity, medication adherence, exacerbation adherence), predisposing behavior change outcomes (self-efficacy, knowledge, self-determination theory constructs), and clinical outcomes (quality of life, exercise tolerance) between the Traditional PR group compared to the new Canadian Standardized PR group.

Patients' adherence to action plan and regular medication, self-efficacy, symptoms/health: After carefully examining data for distribution (and transforming if warranted), the investigators will first calculate the proportion (and 95% CI) of patients who initiate their action plan, including seeking treatment and increasing medications as appropriate within 48 hours of symptom onset. In the case of multiple exacerbations, only the first instance will be used. A separate analysis will be done for multiple exacerbations, to account for patient variables. The investigators will explore secondary objectives by evaluating changes over time in all patients in adherence to medication, self-efficacy, symptoms and, health related quality of life. Regression analyses will be used to explore changes in these outcomes while controlling for the effects of potential covariates and confounders such as baseline respiratory status, age, sex, disease severity, comorbidities and smoking status. The investigators will calculate means or proportions for acceptability to providers and resource use.

Sample Size Determination: The investigators anticipate a sample of 200 COPD patients (100 in each group), with 40 of those patients participating in rural sites by Tele-health. Sample size calculations are based on evaluating change in the primary outcome - physical activity as measured by steps per day - between the Traditional PR and new Canadian Standardized PR groups. A literature search indicated that Traditional PR seems to have a small to negligible effect on COPD patients' physical activity levels. Given that the new Canadian Standardized program is designed to specifically target predisposing factors of behavior change, the investigators anticipate a medium effect size increase in physical activity compared to the usual care program. In order to detect a medium effect size, with power = .80, and alpha = .05, the investigators will be recruiting 100 COPD patients per group (G*Power 3).

Data Handling and Record Keeping: Data will be collected and stored in a central Redcap database. Patients will all have a unique study code number, which will be the only unique identifier included within the Redcap database.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be enrolled into pulmonary rehabilitation within our affiliated PR sites, or in satellite Tele-health program, with a diagnosis of COPD confirmed by post-bronchodilator forced expiratory volume in 1 second by forced vital capacity (FEV1/FVC) ratio of less than 0.7.
* Patients must be able to read and communicate in English or French.

Exclusion Criteria:

* Patients enrolled into pulmonary rehabilitation with a diagnosis other than COPD will be excluded.
* Patients with cognitive impairments who are unable to accurately complete questionnaires will also be excluded.
* As part of standard rehabilitation referral procedures, all patients must be ambulatory and not have unstable cardiovascular disease.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Physical activity assessed as steps per day as evaluated by Fitbit | Change from baseline physical activity to the end of rehabilitation (6-8 weeks) and 6 months post-rehabilitation

SECONDARY OUTCOMES:
Patient adherence to exacerbation action plan | 6 months after rehabilitation has ended
Medication adherence assessed by pharmacy refill records | 6 months after rehabilitation has ended

OTHER OUTCOMES:
Multidimensional Self-efficacy for Exercise Scale | Change from baseline to the end of rehabilitation (6-8 weeks) and 6 months post-rehabilitation
Self-efficacy for Walking Scale | Change from baseline to the end of rehabilitation (6-8 weeks) and 6 months post-rehabilitation
Self-efficacy for Medication Adherence | Change from baseline to the end of rehabilitation (6-8 weeks) and 6 months post-rehabilitation
COPD Knowledge | Change from baseline to the end of rehabilitation (6-8 weeks), and 6 months post-rehabilitation
Psychological Need Satisfaction for Exercise Scale | Change from baseline to the end of rehabilitation (6-8 weeks) and 6 months post-rehabilitation
Psychological Need Thwarting Scale | Change from the end of rehabilitation (6-8 weeks) to 6 months after rehabilitation
Treatment Self-regulation Questionnaire | Change from baseline to the end of rehabilitation (6-8 weeks) and 6 months post-rehabilitation
Functional exercise capacity assessed by the 6-minute walk test | Change from baseline to the end of rehabilitation (6-8 weeks) and 6 months post-rehabilitation
Health-related quality of life assessed by the COPD Assessment Tool | Change from baseline to the end of rehabilitation (6-8 weeks) and 6 months post-rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Michael K Stickland, PhD, Principal Investigator — University of Alberta
Locations (1):
- G. F. MacDonald Centre for Lung Health, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Selzler AM, Jourdain T, Wald J, Sedeno M, Janaudis-Ferreira T, Goldstein R, Bourbeau J, Stickland MK. Evaluation of an Enhanced Pulmonary Rehabilitation Program: A Randomized Controlled Trial. Ann Am Thorac Soc. 2021 Oct;18(10):1650-1660. doi: 10.1513/AnnalsATS.202009-1160OC. PMID 34004123